CLINICAL TRIAL: NCT05121740
Title: Extension Study in a Cohort of Adult Patients With SARS-CoV-2 Infection Requiring Hospital Admission and Received Treatment With Plitidepsin in the APLICOV-PC Study
Brief Title: Extension Study in a Cohort of Adult Patients With COVID-19 Infection
Acronym: E-APLICOV-PC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PharmaMar (Industry)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-APL-A-003-21; 2021-004966-37 (EudraCT Number)
Record Dates: First submitted 2021-11-08; First posted 2021-11-16 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: COVID-19 Infection
Keywords: Plitidepsin; COVID-19; Post-COVID morbidity
MeSH Terms: conditions — COVID-19 | interventions — plitidepsin

STUDY DESIGN:
Intervention Model Description: Follow up Multicentric extension study of APLICOV-PC clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: Experimental 1 (Experimental): In the APLICOV-PC study, patients of arm A received 1.5 mg of plitidepsin / day for 3 consecutive days (total dose 4.5 mg).
  Interventions: Drug: Plitidepsin 1.5 mg / day
- Arm B: Experimental 2 (Experimental): In the APLICOV-PC study, patients of arm B received 2.0 mg of plitidepsin / day for 3 consecutive days (total dose 6.0 mg).
  Interventions: Drug: Plitidepsin 2.0 mg / day
- Arm C: Experimental 3 (Experimental): In the APLICOV-PC study, patients of arm C received 2.5 mg of plitidepsin / day for 3 consecutive days (total dose 7.5 mg).
  Interventions: Drug: Plitidepsin 2.5 mg / day

INTERVENTIONS:
Drug: Plitidepsin 1.5 mg / day — Plitidepsin 1.5 mg/day infused through a pump device over 1 hour and 30 minutes, 3 consecutive days (total dose 4.5 mg).
  Arms: Arm A: Experimental 1
Drug: Plitidepsin 2.0 mg / day — Plitidepsin 2.0 mg/day infused through a pump device over 1 hour and 30 minutes, 3 consecutive days (total dose 6.0 mg).
  Arms: Arm B: Experimental 2
Drug: Plitidepsin 2.5 mg / day — Plitidepsin 2.5 mg/day infused through a pump device over 1 hour and 30 minutes, 3 consecutive days (total dose 7.5 mg).
  Arms: Arm C: Experimental 3

SUMMARY:
The main objective of this study is to evaluate the incidence of post-COVID morbidity and characterize the complications profile in patients who participated in the APLICOV-PC study. APLICOV-PC study was a multicenter, randomized, proof-of-concept clinical trial to assess the safety profile of 3 different dose levels of plitidepsin (1,5 mg, 2,0 mg and 2,5 mg) administered three consecutive days, in adult patients with confirmed diagnosis of COVID-19 who require hospital admission.

DETAILED DESCRIPTION:
The APLICOV-PC proof of concept study demonstrated the antiviral activity of plitidepsin in terms of reducing viral load, inducing recovery, and impact on lymphocyte reconstitution and other inflammatory parameters.

A percentage of patients, which varies between 10 and 25%, continue to show symptoms at 3 months after contracting the Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection: For some of them this significantly restricts their life, requiring them to take long-term sickness leave from work, and leaving them with sequelae that may continue for more than one year.

With this study, Pharmamar intends to evaluate whether the treatment with plitidepsin, by attaining a reduction in the viral load and a faster recovery of the patient, could have a relevant impact on the emergence of sequelae resulting from the SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient who participated in the APLICOV-PC study receiving treatment with plitidepsin and who gives consent.

Exclusion Criteria:

* There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José Felipe Varona, MD, Principal Investigator — Hospital Universitario HM Montepríncipe; Pedro Landete, MD, Principal Investigator — Hospital Universitario La Princesa; Pablo Guisado-Vasco, MD, Principal Investigator — Quironsalud; Roger Paredes, MD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (10):
- Spain (10):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario HM Montepríncipe, Boadilla del Monte, Madrid
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital Universitario de Getafe, Getafe
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid

REFERENCES:
- [Background] Varona JF, Landete P, Paredes R, Vates R, Torralba M, Guisado-Vasco P, Porras L, Munoz P, Gijon P, Ancochea J, Saiz E, Meira F, Jimeno JM, Lopez-Martin JA, Estrada V. Plitidepsin in adult patients with COVID-19 requiring hospital admission: A long-term follow-up analysis. Front Cell Infect Microbiol. 2023 Feb 22;13:1097809. doi: 10.3389/fcimb.2023.1097809. eCollection 2023. PMID 36909731
- See also: Related Info — http://www.frontiersin.org/articles/10.3389/fcimb.2023.1097809/full

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were included in the study between 25th January 2022 and 28th February 2022.
Pre-assignment Details: All patients who participated in and received plitidepsin in the APLICOV-PC study are eligible candidates for participating in this extension study.
Groups:
- Arm A: Experimental 1: 1.5 mg of plitidepsin / day
- Arm B: Experimental 2: 2.0 mg of plitidepsin / day
- Arm C: Experimental 3: 2.5 mg of plitidepsin / day
Period: Overall Study
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3
Started | 9 | 14 | 11
Completed | 9 | 14 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Age, Continuous [Median (Full Range); unit: years] | 53 [33 to 70] | 52.5 [36 to 72] | 54 [43 to 68] | 53 [33 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 11
  Male | 7 | 10 | 6 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 7 | 9 | 7 | 23
  Latin | 2 | 3 | 4 | 9
  North African | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1
Weight [Median (Full Range); unit: Kg] | 80.0 [50 to 106] | 88.5 [62 to 140] | 86.0 [54 to 145] | 84.8 [50 to 145]
Height [Median (Full Range); unit: cm] | 170.0 [160 to 182] | 169.0 [148 to 187] | 161.0 [152 to 187] | 168.4 [148 to 187]
Body Surface Area [Median (Full Range); unit: m^2] | 1.9 [1.5 to 2.2] | 2.0 [1.6 to 2.5] | 1.9 [1.5 to 2.6] | 1.9 [1.5 to 2.6]

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Complications Related to Post COVID-19 Infection
Description: Number and percentage of patients who developed complications related to post COVID-19 infection
Time Frame: Since last visit of APLICOV-PC study until the end of this extension study, an average of 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Participants | 4 | 8 | 5 | 17

2. Secondary Outcome: Patients Requiring Oxygen Therapy
Description: Percentage of patients requiring oxygen therapy
Time Frame: Since last visit of APLICOV-PC study until the end of this extension study, an average of 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Participants | 1 | 2 | 0 | 3

3. Secondary Outcome: Patients With Complications Post COVID-19 Infection (Regardless Relationship, i.e. Related to COVID-19 Infection or Not).
Description: Percentage of patients with complications Post COVID-19 Infection (Regardless Relationship, i.e. Related to COVID-19 Infection or Not).
Time Frame: Since last visit of APLICOV-PC study until the end of this extension study, an average of 12 months..
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Participants
  Without complications | 1 | 2 | 5 | 8
  Regardless relationship, i.e. related to COVID-19 infection or not. | 8 | 12 | 6 | 26

4. Secondary Outcome: Ratio of Partial Pressure Arterial Oxygen (PaO2) and Fraction of Inspired Oxygen (FiO2)
Description: PaO2/FiO2 (Ratio of partial pressure arterial oxygen and fraction of inspired oxygen) mean, standard deviation.
  PaO2/FiO2 ratio to evaluate disease severity and discriminate between 'Moderate' and 'Severe' categories according to FDA guidance.
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Ratio | 472.0 (85.9) | 464.2 (90.3) | 518.7 (99.1) | 482.8 (92.2)

5. Secondary Outcome: Forced Expiratory Volume 1 (FEV1)
Description: FEV1 (Forced expiratory volume 1) mean, standard deviation.
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
ml | 3052 (865.4) | 3267 (774.9) | 2857 (1029) | 3078 (877.9)

6. Secondary Outcome: Lung Diffusion Testing
Description: Lung difussion testing: mean and standard deviation. Unit of measure: % reference theoretical value
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Mean (Standard Deviation); unit: Percentage reference theoretical value
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Percentage reference theoretical value | 98.4 (11.4) | 100.1 (24.0) | 105.2 (15.2) | 101.3 (18.4)

7. Secondary Outcome: Patients With Alterations in Chest Radiography
Description: Percentage of patients with alterations in chest radiography
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Patients With Electrocardiogram Alterations
Description: Percentage of patients with electrocardiogram alterations
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Participants | 1 | 3 | 1 | 5

9. Secondary Outcome: Patients With ≥Grade 2 Alterations in Laboratory Parameters
Description: Percentage of patients with ≥grade 2 alterations in laboratory parameters Grade measured according to NCI-CTCAE v5.0 (National Cancer Institute - Common Terminology Criteria for Adverse Events version 5.0) where Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL* Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Participants | 1 | 1 | 1 | 3

10. Secondary Outcome: Modified Medical Research Council (mMRC) Dyspnea Scale
Description: Percentage of patients in each category of the Modified Medical Research Council (mMRC) dyspnea scale.
  The mMRC scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4:
  0, no breathlessness except on strenuous exercise;
  1. shortness of breath when hurrying on the level or walking up a slight hill;
  2. walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level;
  3. stops for breath after walking ∼100 m or after few minutes on the level; and
  4. too breathless to leave the house, or breathless when dressing or undressing.
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Participants
  0 | 5 | 7 | 9 | 21
  1 | 2 | 6 | 2 | 10
  2 | 0 | 1 | 0 | 1
  3 | 2 | 0 | 0 | 2

11. Secondary Outcome: FEV1/FVC
Description: FEV1/FVC mean, standard deviation.
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Ratio | 79.9 (5.8) | 79.3 (8.6) | 78.1 (13.0) | 79.1 (9.4)

12. Secondary Outcome: Forced Vital Capacity (FVC)
Description: FVC mean, standard deviation.
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
ml | 3809 (1022) | 4107 (827.2) | 3751 (1222) | 3913 (1001)

13. Secondary Outcome: Arterial Oxygen Saturation (SaO2)
Description: SaO2 (Arterial oxygen saturation) mean, standard deviation. Unit of measure: percentage of oxygen saturation
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Percentage of oxygen saturation | 97.2 (1.8) | 97.1 (1.7) | 98.1 (1.2) | 97.4 (1.6)

14. Secondary Outcome: Barthel Index
Description: The Barthel index measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL) i.e. feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing.
  Percentage of patients at each category according to the score obtained: 0-20: Total dependence; 21-60: Severe dependence; 61-90: Moderate dependence; 91-99: Low dependence; 100: Independence
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Participants
  Obtained | 0 | 0 | 0 | 0
  Total dependence | 0 | 0 | 0 | 0
  Severe dependence | 0 | 0 | 0 | 0
  Moderate dependence | 0 | 0 | 0 | 0
  Low dependence | 0 | 0 | 0 | 0
  Independence | 9 | 14 | 11 | 34

15. Secondary Outcome: Patients Requiring Hospital Readmission
Description: Percentage of patients requiring hospital readmission
Time Frame: Since last visit of APLICOV-PC study until the end of this extension study, an average of 12 months.
Measure: Count of Participants; unit: Participants
Groups:
- Total: No applicable
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Participants
  Post-COVID-19 complications | 0 | 0 | 0 | 0
  COVID-19 | 0 | 0 | 0 | 0
  No COVID-19 related | 0 | 1 | 0 | 1
  No readmission | 9 | 13 | 11 | 33

16. Secondary Outcome: 6 Minute Walking Test (Total Distance)
Description: minute walking test mean, standard deviation. Total distance measured in meters (m)
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
m | 486.4 (115.8) | 453.9 (77.7) | 445.1 (134.0) | 459.7 (106.5)

17. Secondary Outcome: 6 Minute Walking Test (Expected Distance)
Description: minute walking test mean, standard deviation. Expected distance (the predicted distance that a patient could walk) measured in meters (m)
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
m | 806.7 (101.7) | 853.5 (149.7) | 818.7 (101.9) | 829.8 (122.1)

18. Secondary Outcome: 6 Minute Walking Test (Percentage of Predicted Distance)
Description: 6 minute walking test mean, standard deviation. Unit of measure: Percentage of predicted distance
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Mean (Standard Deviation); unit: Percentage of predicted distance
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Percentage of predicted distance | 61.4 (16.8) | 54.3 (11.9) | 54.6 (16.6) | 56.3 (14.8)

19. Secondary Outcome: 6 Minute Walking Test (Number of Laps of 60 m)
Description: 6 minute walking test mean, standard deviation. Unit of measure: Number of laps of 60 m
Time Frame: At study inclusion, an average of 12 months after end of APLICOV-PC study.
Measure: Mean (Standard Deviation); unit: Number of laps of 60 m
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3 | Total
Number analyzed (Participants) | 9 | 14 | 11 | 34
Number of laps of 60 m | 22.8 (14.7) | 14.0 (7.2) | 15.7 (12.5) | 16.9 (11.6)

ADVERSE EVENTS:
Time Frame: From the informed consent signature to the end of study, approximately 1 month
Description: No adverse events were reported during study period.
Groups:
- Arm B: Experimental 2: 2.0 mg of plitidepsin / day f
Arm/Group | Arm A: Experimental 1 | Arm B: Experimental 2 | Arm C: Experimental 3
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/14 | 0/11

LIMITATIONS AND CAVEATS:
Low sample size and a lack of control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT05121740/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT05121740/SAP_001.pdf